CLINICAL TRIAL: NCT04072991
Title: E-C DIBS: Randomised Controlled Study: Comparing the Effectiveness and Convenience of Dietary Therapy for Irritable Bowel Syndrome (IBS)
Brief Title: A Study Comparing the Effectiveness and Convenience of Dietary Therapy for Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH20655
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low FODMAP diet (Active Comparator): As part of their treatment for IBS participants may be randomised to a low FODMAP diet
  Interventions: Other: dietary therapy
- Gluten Free Diet (Active Comparator): As part of their treatment for IBS participants may be randomised to a gluten free diet
  Interventions: Other: dietary therapy
- British Dietetic Association diet (Active Comparator): As part of their treatment for IBS participants may be randomised to the BDA diet
  Interventions: Other: dietary therapy

INTERVENTIONS:
Other: dietary therapy — participants will undertake a four week diet as part of their IBS treatment

SUMMARY:
Irritable bowel syndrome is a functional lower gastrointestinal disorder characterised by abdominal pain and altered bowel habit in the absence of organic pathology to explain the symptoms. Irritable bowel syndrome has a prevalence of approximately 10% in adults, shows a female preponderance, and is more common in younger individuals. In clinical practice, Irritable bowel syndrome accounts for almost a third of all gastroenterology cases seen in primary care, with a subsequent third of these being referred onto secondary-care for further evaluation. The economic burden of Irritable bowel syndrome, in terms of medical expense, work absenteeism and loss of productivity, is considerable.

The exact cause of irritable bowel syndrome is unknown. Accordingly there has been a huge surge in interest for dietary therapies to help manage Irritable bowel syndrome. To date, there are only a handful of small randomized controlled trials evaluating the efficacy of dietary therapy in Irritable bowel syndrome. In light of this we plan to conduct the first randomized controlled trial directly comparing the effectiveness of the low-FODMAP diet, British Dietetic Association diet, and the gluten free diet in Irritable bowel syndrome. Moreover, such a trial allows for a direct comparison of nutritional and gut microbial changes, both of which can suffer detrimental consequences following the implementation of restrictive dietary therapies. This study is also unique in that it takes into consideration the patients' perspective with regards to the convenience and cost-effectiveness of implementing such diets into routine day-to-day life. The study will aim to recruit 100 patients from Sheffield Teaching Hospitals gastrointestinal clinics. Following recruitment patients will be seen by a hospital dietitian where they will be randomized to one of the 3 diets. Participants will complete a questionnaire portfolio weekly for one month as part of the study

ELIGIBILITY:
Inclusion Criteria:

1. Irritable Bowel syndrome - as defined by abdominal pain and altered bowel habit in the absence of organic pathology to explain the symptoms.This is the contemporary definition as provided by the Rome IV committee.
2. Age 18-65 years
3. English literate
4. Can travel to hospital
5. Telephone/internet access

Exclusion Criteria:

1. Inflammatory bowel disease
2. Coeliac disease
3. Gastrointestinal cancer
4. Previous abdominal surgery
5. Scleroderma
6. Poorly controlled diabetes
7. Severe liver disease
8. Severe renal disease
9. Severe respiratory disease
10. Severe cardiac disease
11. Severe psychiatric disease
12. Memory disorders
13. Pregnant
14. Current dietary interventions
15. Recent/current use of Probiotics
16. Recent/current use of Antibiotics
17. Recent/current use of Narcotics
18. Currently titrated antidepressants (i.e. not on a stable dose)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage with at least 50-point reduction in Irritable bowel syndrome Severity Scoring System questionnaire | Baseline to week 4
  A validated questionnaire to assess IBS symptoms and severity. The ranges of this questionnaire are included below:
  How severe was your pain? 0 (no pain) -100 (very severe)
  how severe is your abdominal (tummy) pain? 0 (no pain) - 100 (very severe)
  how severe is your abdominal distention/tightness? 0 (no pain) - 100 (very severe)
  How satisfied are you with your bowel habit? 0 (very happy) - 100 (very unhappy)
  Please indicate with a cross on the line below how much your irritable bowel syndrome is affecting or interfering with your life in general. 0 (not at all) - 100 (completely)
  A higher score on any scale represents a negative outcome.
  A ≥ 50-point reduction in IBS-SSS following intervention represents a clinically significant improvement

SECONDARY OUTCOMES:
Changes in proportion with anxiety and depression | Baseline to week 4
  Hospital Anxiety and Depression Scale - is a psychological screening tool to which there are in total 14 items, seven each for depression and anxiety. Each item is rated from 0 (not present) to 3 (maximum), giving a cumulative score for each subscale to range from 0 to 21. A subscale score of ≥11 is used to indicate a clinically significant level of anxiety or depression.
Changes in somatization | Baseline to week 4
  The patient health questionnaire (PHQ)-12 non-GI somatic symptoms scale- The PHQ-12 records bothersome non-GI symptoms over the past month. The twelve symptoms assessed are back pain, limb pain, headaches, chest pain, dizziness, fainting spells, palpitations, breathlessness, menstrual cramps, dyspareunia, insomnia, and lethargy. Subjects were asked to rate how much they had been troubled by these 12 symptoms over the last four weeks as 0 ("not bothered at all"), 1 ("bothered a little"), or 2 ("bothered a lot"). Responses were used to calculate the number of sites reporting somatic symptoms (ranging from 0 to 12) and the somatisation severity score (ranging from 0 to 24), which was categorised as minimal (less than or equal to 3), low (4-7), medium (8-12) and high (≥ 13).
Changes in IBS-quality of life | Baseline to week 4
  The IBS quality of life (IBS-QOL) questionnaire - this consists of 34 questions which are summed and averaged for a total score, in addition to eight subscale scores (Dysphoria, Interference with Activity, Body Image, Health Worries, Food Avoidance, Social Reaction, Sexuality, Social Relationship). Total and subscale scores are transformed to a 0-100 scale. Higher scores indicate better IBS-specific QOL.
Acceptability of dietary restriction | Week 4
  The acceptability of dietary restriction questionnaire is based on the adapted nutrition related quality of life (QOL) questionnaire. Responses are recorded using a Likert scale, with the responses of agree, neutral and disagree.
Food related quality of life (QOL) questionnaire | Week 4
  The food related QOL questionnaire is a seven-item questionnaire based on the food-related QOL tool (Satisfaction with Food-related Life). Responses are recorded on Likert scale, as either agree, neutral and disagree.
Comprehensive Nutrition Assessment Questionnaire | Baseline to week 4
  The Comprehensive Nutrition Assessment Questionnaire is a semi-quantitative food frequency questionnaire, consisting of 297 questions, assessing macronutrient and micronutrient intake, as well as FODMAPs, fibre, starch, glycaemic index and glycaemic load
Changes in stool dysbiosis index | Baseline to week 4
  Participants will provide a stool sample both pre- and post-dietary intervention. Data will be analysed by using the GA-map™ Dysbiosis Test (Genetic Analysis AS, Oslo, Norway). Bacterial profiles will be assigned a dysbiosis index (DI), on a scale from 0 to 5, with a DI score of 2 or lower being classified as being within the non dysbiotic region compared to the normobiotic reference range. A DI score of greater than 2 will be considered to be dysbiotic, with a higher DI number indicating greater dysbiosis from the reference range.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Aziz, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] Rej A, Sanders DS, Shaw CC, Buckle R, Trott N, Agrawal A, Aziz I. Efficacy and Acceptability of Dietary Therapies in Non-Constipated Irritable Bowel Syndrome: A Randomized Trial of Traditional Dietary Advice, the Low FODMAP Diet, and the Gluten-Free Diet. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2876-2887.e15. doi: 10.1016/j.cgh.2022.02.045. Epub 2022 Feb 28. PMID 35240330